CLINICAL TRIAL: NCT07051408
Title: Predictors Of Cognitive Decline In Attenders Of Essex Memory Clinic From Digital Devices Using Classical Statistical Methods, Machine Learning And Disease Progression Modelling
Brief Title: Predictors Of Cognitive Decline Using Digital Devices
Acronym: CODEC-II
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 144168; IRAS ID: 289028 (Other: Health Research Authority)
Record Dates: First submitted 2025-06-17; First posted 2025-07-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD); Rapid Eye Movement Sleep Behavior Disorder; Healthy Control Patients of the Same Age
Keywords: Digital Devices; Diagnosis; Prediction; Prognosis; Dementia Risk; Machine Learning; Wearables; Blood Based Biomarkers
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; REM Sleep Behavior Disorder; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, Cellular Fraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this study is to find out if people with cognitive difficulties will wear and use different types of digital technology, and if they will allow data from that technology and their clinical profile to be collected. Participants will be patients in Essex Memory clinic and their partners/carers. The digital technology used will include a smartwatch, a sleep headband and two smartphone applications, which have been selected as part of the Early Detection of Neurodegenerative Disease (EDoN) initiative. The investigators will also investigate how the digital data can be analyzed together with routinely captured clinical data using machine learning models, a complex type of statistical analysis.

The aim of the wider EDoN initiative is to combine digital and clinical data to develop machine learning models which can predict individuals' risk of developing dementia decades before the onset of symptoms.

DETAILED DESCRIPTION:
Study Design & Methods of Data Collection: This study is designed as an observational, pilot and feasibility study. Recruitment will be over 18 months with clinical data collected at baseline and up to 5 years follow up, and digital data collected at baseline, 3, 6, 9 and 12 months.

Setting: Essex Memory Clinics within the Essex Partnership University NHS Foundation Trust which serves older adults living in greater London and Essex areas.

Participants: The investigators aim to recruit a minimum of 100 participants, comprising of a 3:1 ratio of patients to controls respectively (refer to section 6 for eligibility criteria). Participants will include patients of the memory clinic with cognitive complaints, mild cognitive impairment or dementia, and their partners/carers/family members/friends as controls. As this is a feasibility study, this sample is not based on a power calculation, but findings will inform future work in this area. Sampling will follow a convenience strategy, appropriate for a feasibility study.

Methods: Overall feasibility of implementing digital tools within a clinical population will be evaluated through a combination of direct usage data from the devices and apps and via questionnaires. Digital tools (Fitbit, Dreem headband, Mezurio app, Longevity app) will be provided to participants at a baseline visit at the participant's home.

The broad, but not exclusive, areas of interest will include:

* Participant retention and attrition rates of each digital tool
* Comparison of 14- and 28-day Mezurio schedules
* Practicalities of distribution, collection and storage of the digital technologies
* Approaches to train participants on use of digital technologies
* Technical support needs and uptake by participants
* Ease of transfer and integration of digital data
* Assessment of the study management platform (Fluvial)

Digital Tools: In order to develop disease-specific fingerprint models, it is necessary to collect a wide range of measures which may be affected by early disease processes. Therefore, a combination of digital tools will be utilised, including remote active and passive smartphone-based assessments and remote passive data collection with devices (e.g., a smartwatch and an EEG headband). These technologies will be targeted at functions with a direct relationship to the brain-regions first affected by dementia-related pathology in addition to using digital devices to measure new signals of interest. The investigators will aim to keep the participant burden as low as possible by mainly including passive measures (e.g., monitoring sleep EEG) and by limiting the amount of time participants are engaged in active assessments (e.g., a smartphone-based memory test) to approximately 10 minutes per day.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who present to the Essex Memory Clinic and their relatives or carers
2. Capacity to provide written informed consent
3. Sufficient proficiency in English to understand study documents and use the digital devices
4. Own a compatible smartphone (Android 7.0 or higher / iOS 12.2 or higher). If participants own a smartphone which is not a compatible device (i.e. prior to Android 7.0 or iOS 12.2), a new handset will be provided to them, as long as they are willing to use this as their primary phone.
5. Ability to use a smartphone and EDoN digital devices, either alone, or with appropriate support (carer, partner, family member, etc). Support would involve reminding participants to complete study tasks and to charge / wear devices.
6. Able to connect to the internet using their smartphone at home. Note: In order to use the Dreem headband, participants will additionally require a home WiFi connection. However, participants without a WiFi connection will still be able to join the study and will not be asked to use the Dreem headband.
7. For people with a diagnosis of dementia, a carer, partner or family member willing to support their participation in the study by reminding patients to complete study tasks and to charge/wear their devices
8. For patients who do not have a record of neurocognitive and physical assessments outlined in section 4.5.3, they must be willing to undergo these additional assessments
9. For the blood donation sub study only: consented to participate in the main CODEC II study.
10. For the qualitative sub study only: able to use a phone or video-conferencing platform to participate in the interviews
11. Aged 40+ years

Exclusion Criteria:

1. Patients with active major psychiatric disorder which requires regular reviews by secondary care, for example schizophrenia, schizoaffective disorder or bipolar affective disorder
2. Patients under end-of-life care
3. Previous sensitivity or allergic skin reaction to latex, rubber or plastics
4. Do not have a personal smartphone with internet access
5. Participating in a clinical trial of an investigational medicinal product
6. Not meeting all inclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include patients of Essex Memory Clinics within the Essex Partnership University NHS Foundation Trust which serves older adults living in greater London and Essex areas. Participants will be patients with cognitive complaints, mild cognitive impairment or dementia, and their partners/carers/family members/friends as controls.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean proportion (%) of scheduled digital data capture visits fully completed for each digital technology (Fitbit Charge 4/5, Dreem 2/3 headband, Mezurio smartphone app, and Longevity smartphone app) at each timepoint | 0, 3, 6, 9, and 12 months
  The investigators will assess the feasibility of capturing digital data from digital technologies that have been selected as part of the EDoN initiative. This will be achieved by assessing the mean proportion (%) of scheduled digital data capture visits fully completed for each digital technology (Fitbit Charge 4/5, Dreem 2/3 headband, Mezurio smartphone app, and Longevity smartphone app) at each timepoint. In addition, a subset of participants who consented to the main study will be invited to participate in a qualitative sub-study to explore the perspectives of people with cognitive impairment and their partners, carers or family members on the use of digital devices included in the EDoN toolkit.
Mean proportion (%) of scheduled Mezurio data capture visits fully completed at each timepoint for individuals randomised to 14- and 28-day Mezurio schedules | 0, 3, 6, 9, and 12 months
  One of the digital technologies being evaluated/utilised in the study is a cognitive testing application called 'Mezurio' created by Dr Chris Hinds at the University of Oxford. Participants will be asked to install Mezurio on their smartphone at baseline and complete a range of short tasks over a period of either 14 or 28 consecutive days during the 12 month study period. Participants on the 14 day schedule will repeat the assessments at 3 month intervals; participants on the 28 day schedule will repeat the assessments at 6 month intervals. Participants will be allocated to each assessment period randomly. The investigators will assess the mean proportion (%) of scheduled Mezurio data capture visits fully completed at each timepoint for individuals randomised to 14- and 28-day Mezurio schedules.

SECONDARY OUTCOMES:
Incident subjective cognitive decline (SCD), mild cognitive impairment (MCI), or dementia | 12 months
  In participants who are patients (recruited from memory clinics), the investigators will record new diagnoses that represent a progression/worsening of cognitive decline. For example, in patients with SCD, the investigators will record incident MCI/dementia, whereas for patients with MCI, only incident dementia will be recorded.
  In participants who are relatives/carers (i.e., healthy controls), the investigators will record any new cognitive diagnoses, including SCD, MCI and/or dementia. These data will be used to achieve the broader aims of the study (please see Study Description for details).

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Walker, MD, Principal Investigator — University College, London
Locations (1):
- St Margarets Hospital, Epping, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Digital device data, demographic data and some clinical data.
Time Frame: Q1 2027 for five years
Access Criteria: Bona fide researchers
URL: https://www.alzheimersdata.org/ad-workbench

REFERENCES:
- [Derived] Wilson S, Beswick E, Morrell R, Bhogal S, Tolley C, Whitfield T, Wing K, Mc Ardle R, Hassan N, Walker Z, Slight S. Acceptability of wearable technology for the early detection of dementia-causing diseases: perspectives from the CODEC II cohort. BMC Digit Health. 2025;3(1):55. doi: 10.1186/s44247-025-00191-3. Epub 2025 Aug 29. PMID 40893385